CLINICAL TRIAL: NCT00111631
Title: A Randomized, Double-blind Study of the Effect of the DPP-IV Inhibitor on HbA1c and Safety in Patients With Type 2 Diabetes Treated With a Stable Dose of Metformin
Brief Title: A Study of DPP-IV Inhibitor in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM18106
Record Dates: First submitted 2005-05-24; First posted 2005-05-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dipeptidyl-Peptidase IV Inhibitors; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: DPP-IV Inhibitor; Drug: Metformin
- 2 (Experimental)
  Interventions: Drug: DPP-IV Inhibitor; Drug: Metformin
- 3 (Experimental)
  Interventions: Drug: DPP-IV Inhibitor; Drug: Metformin
- 4 (Placebo Comparator)
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: DPP-IV Inhibitor — Escalating doses po bid
  Arms: 1; 2; 3
Drug: Metformin — As prescribed
Drug: Placebo — po bid
  Arms: 4

SUMMARY:
This study will assess the efficacy, safety and tolerability of DPP-IV Inhibitor in patients with type 2 diabetes receiving a stable dose of metformin. The anticipated time on study treatment is 3-12 months and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-75 years of age;
* type 2 diabetes;
* stable metformin therapy for >=3 months before screening.

Exclusion Criteria:

* women who are pregnant, breast-feeding, or not using an adequate contraceptive method;
* type 1 diabetes;
* any anti-hyperglycemic medication other than metformin in the last 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2005-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in HbAlc\n | Week 16

SECONDARY OUTCOMES:
Absolute change in FPG and absolute/relative change in insulin sensitivity, beta-cell-function, and lipid profile, response rate\n | Week 16
AEs, vital signs, laboratory tests, body weight, waist/hip ratio, ECG\n | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- United States (20):
  - Concord, California
  - Salinas, California
  - San Diego, California
  - Boulder, Colorado
  - Newark, Delaware
  - Wilmington, Delaware
  - Clearwater, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Detroit, Michigan
  - Buffalo, New York
  - Rochester, New York
  - Durham, North Carolina
  - Mogadore, Ohio
  - Portland, Oregon
  - Connellsville, Pennsylvania
  - Warminster, Pennsylvania
  - Dallas, Texas
  - Midland, Texas
  - San Antonio, Texas
- Australia (2):
  - Adelaide
  - Sydney
- Canada (4):
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - London, Ontario
  - Toronto, Ontario
- Germany (6):
  - Bad Lauterberg im Harz
  - Berlin
  - Dresden
  - Görlitz
  - Mainz
  - Neuss
- Italy (4):
  - Ancona
  - Florence
  - Napoli
  - Udine
- Ponce, Puerto Rico